CLINICAL TRIAL: NCT04225078
Title: A Randomized, Double-blind, Placebo- and Positive-controlled, Single-dose, 4 Way Crossover Study to Evaluate the Effects of Loperamide (JNJ-289679) on Electrocardiogram Intervals in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effects of Loperamide (JNJ-289679) on Electrocardiogram Intervals in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CR108643; 2019-003776-39 (EudraCT Number); R018553NAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Loperamide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: Treatment ADBC (Experimental): Participants will receive treatment A (Loperamide therapeutic dose) on Day 1 on treatment period 1, followed by Treatment D (Moxifloxacin) on Day 1 of treatment period 2 followed by Treatment B (Loperamide supratherapeutic dose) on Day 1 of treatment period 3 followed by Treatment C (placebo) on Day 1 of treatment period 4. Each treatment period will be separated by a minimum of 7-day washout period and no more than 21-day.
  Interventions: Drug: Loperamide; Other: Placebo; Drug: Moxifloxacin
- Treatment Sequence 2: Treatment BACD (Experimental): Participants will receive Treatment B on Day 1 of treatment period 1 followed by Treatment A on Day 1 of treatment period 2 then Treatment C on Day 1 of treatment period 3 and then Treatment D on Day 1 of treatment period 4. Each treatment period will be separated by a minimum of 7-day washout period and no more than 21-day.
  Interventions: Drug: Loperamide; Other: Placebo; Drug: Moxifloxacin
- Treatment Sequence 3: Treatment CBDA (Experimental): Participants will receive Treatment C on Day 1 of treatment period 1 followed by Treatment B on Day 1 of treatment period 2 then Treatment D on Day 1 of treatment period 3 and then Treatment A on Day 1 of treatment period 4. Each treatment period will be separated by a minimum of 7-day washout period and no more than 21-day.
  Interventions: Drug: Loperamide; Other: Placebo; Drug: Moxifloxacin
- Treatment Sequence 1: Treatment DCAB (Experimental): Participants will receive Treatment D on Day 1 of treatment period 1 followed by Treatment C on Day 1 of treatment period 2 then Treatment A on Day 1 of treatment period 3 and then Treatment B on Day 1 of treatment period 4. Each treatment period will be separated by a minimum of 7-day washout period and no more than 21-day.
  Interventions: Drug: Loperamide; Other: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Loperamide — Loperamide will be administered as a single oral dose at the expected therapeutic or supratherapeutic doses respectively.
Other: Placebo — Matching loperamide placebo capsules will be administered orally.
Drug: Moxifloxacin — Moxifloxacin tablets will be administered orally.

SUMMARY:
The purpose of this study is to assess the effects of loperamide on QT/ QT interval corrected for heart rate (QTc) intervals and electrocardiogram (ECG) morphology at therapeutic and supratherapeutic exposures in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* All female participants, except if postmenopausal, must have a negative serum beta-human chorionic gonadotropin (beta hCG) pregnancy test at screening and a negative urine pregnancy test on Day 1 of each treatment period
* A female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 1 month after the last study drug administration
* A male participant, who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Must have a body mass index (body mass index [BMI]; weight kilogram per meter per height per square per meter square [kg/height^2 m^2]) between 18.0 and 30.0 kg/m^2 (inclusive) with a body weight not lower than 50 kilogram (kg)
* Must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. Heart rate between 45 and 100 beats per minute (bpm), inclusive

Exclusion Criteria:

* History of or current renal insufficiency (estimated glomerular filtration rate [eGFR] less than (<) 90 milliliter per minute per meter square (mL/min/1.73m^2) based on the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula at screening only)
* Clinically significant abnormal values for hematology, serum chemistry (including thyroid-stimulating hormone [TSH] at screening only) or urinalysis at screening or at admission to the study site, as deemed appropriate by the investigator. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at screening or at admission to the study site as deemed appropriate by the investigator
* Received a known inhibitor of Cytochrome (CY) P3A4, CYP3A4, CYP2C8, or P-glycoprotein (P-gp) activity within 14 days or a period less than 5 times the drugs' half-life; whichever is longer, before the first dose of the study drug is scheduled
* Received a known inducer of CYP3A4 or CYP2C8 activity within 28 days before the first dose of the study drug is scheduled

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in QT Interval Corrected for Heart Rate (QTc) Intervals for Loperamide | Baseline up to 9 weeks
  Change from baseline in QTc intervals for loperamide at therapeutic and supratherapeutic doses will be reported.
Percentage of Participants with Change from Baseline in T-wave Morphology | Up to 9 weeks
  The percentage of participants in each treatment having T-wave morphology changes from baseline that represent the appearance or worsening of the morphological abnormality will be reported.
Percentage of Participants with Occurrence of Abnormal U-wave Morphology | Up to 9 weeks
  The percentage of participants with the occurrence of abnormal U-waves morphology that represent the appearance or worsening of the morphological abnormality will be reported.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Loperamide and its M1 Metabolite | Up to 9 weeks
  Cmax is defined as the maximum observed plasma concentration.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Loperamide and its M1 Metabolite | Up to 9 weeks
  Tmax is defined as the time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve from the Time of Dosing to the Last Measurable Plasma Concentration AUC (0-last) of Loperamide and its M1 Metabolite | Up to 9 weeks
  AUC (0-last) is defined as the area under the plasma concentration-time curve from the time of dosing to the last measurable plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC[0-inifinity]) of Loperamide and M1 Metabolite | Up to 9 weeks
  (AUC[0-inifinity]) is defined as the area under the plasma concentration-time curve from time zero to infinity, calculated as AUClast+Clast/lambda (z), where Clast is the last observed measurable concentration.
Apparent Terminal Elimination Rate Constant Lambda (z) of Loperamide and its M1 Metabolite | Up to 9 weeks
  Lambda (z) is defined as the apparent terminal elimination rate constant, estimated by linear regression using the terminal log-linear phase of the log-transformed concentration versus time curve.
Apparent Elimination Half-Life Associated with the Terminal Slope (t1/2) of Loperamide and M1 Metabolite | Up to 9 weeks
  t1/2 is defined as the apparent elimination half-life associated with the terminal slope lambda (z) of the semilogarithmic drug concentration-time curve.
Metabolite to parent ratio (M/P) for (AUC[0-inifinity]) of Loperamide and M1 Metabolite | Up to 9 weeks
  M/p ratio is defined as metabolite to parent ratio (M/P) for (AUC[0-inifinity]) corrected for molecular weight using the following molecular weights: loperamide 477.045 gram per mol (g/mol), M1 463.018 g/mol.
Relationship Between Systemic Plasma Concentrations of Loperamide and QT/QTc Changes | Up to 9 weeks
  The relationship between systemic plasma concentrations of loperamide and change in QT/QTc will be reported.
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | Up to 9 Weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency